CLINICAL TRIAL: NCT04718597
Title: Lichtenstein or Robotic TAPP Repair of Groin Hernias After Abdominal Prostatectomy: a Single Centre Retrospective Comparative Study
Brief Title: Repair of Groin Hernias After Abdominal Prostatectomy With Robotic TAPP
Acronym: RAPrTAPP
Status: Completed | Type: Observational
Sponsor: Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Principal Investigator, Filip Muysoms, Principal Investigator, Algemeen Ziekenhuis Maria Middelares
Other Study IDs: MMS.2020.067
Record Dates: First submitted 2020-08-26; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Open hernia repair: Patients who underwent inguinal hernia repair via an open Liechtenstein procedure
  Interventions: Procedure: Open inguinal hernia repair
- Robotic assisted hernia repair: Patients who underwent inguinal hernia repair via robotic assisted laparoscopy
  Interventions: Procedure: Robotic assisted inguinal hernia repair

INTERVENTIONS:
Procedure: Robotic assisted inguinal hernia repair — Robotic assisted inguinal hernia repair with DaVinci Xi system instead of open repair
  Groups: Robotic assisted hernia repair
Procedure: Open inguinal hernia repair — Classical approach (open repair)
  Groups: Open hernia repair

SUMMARY:
This retrospective study investigates if robotic assisted groin hernia repair in patients who previously underwent abdominal prostatectomy has an equal or more favorable clinical outcome, compared to open repair in those patients.

DETAILED DESCRIPTION:
In the personal practice of the investigators, there has been a decrease in open groin hernia repair from 17% to 6% since the introduction of robotic assisted surgery. This reflects a change in indication for complex hernias from an open to a minimal invasive approach. One of the typical indications for open approach before adopting the robotic platform were groin hernias after previous abdominal prostatectomy. Since prostatectomy results in scarring of the retropubic area where we need to dissect during MIS groin hernia repair, an open anterior approach is often suggested. With the enhanced view and instrument dexterity of the robotic platform, the investigators have now changed to a minimal invasive approach in these patients.

Therefore, this study will evaluate the clinical outcome after robotic assisted repair of groin hernias in patients who previously underwent an abdominal prostatectomy in comparison to open groin hernia repair.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Underwent uni-or bilateral groin hernia repair in the period March 2015 - March 2020
* Groin hernia repair via robotic assisted laparoscopy or open surgery
* History of abdominal prostatectomy before the groin hernia repair

Exclusion Criteria:

* Age below 18
* Groin hernia repair via conventional laparoscopy
* Groin hernia repair via open surgery other than Liechtenstein method
* Groin hernia repair without mesh placement

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Patients who underwent robotic assisted or open inguinal hernia repair in the period March 2015 - March 2020 and previously underwent an abdominal prostatectomy.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Intra-hospital complications | From admission until hospital discharge, on average 12-24 hours
  Complications during hospital stay according to Clavien-Dindo
Operative time and per-operative complications | During the hernia repair procedure
  Skin-to-skin operating time and complications during the procedure

SECONDARY OUTCOMES:
Early complications at home | Immediately post hospital discharge until 1 month postoperative
  Complications at 1 month follow-up (readmission, seroma, infection) according to Clavien-Dindo

CONTACTS AND LOCATIONS:
Overall Officials: Filip Muysoms, PhD, Principal Investigator — Algemeen Ziekenhuis Maria Middelares
Locations (1):
- AZ Maria Middelares, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: Undecided